CLINICAL TRIAL: NCT01674023
Title: MicroRNA Expression Profile in Human Vitreous of Patients With Various Vitreoretinal Diseases Requiring Vitrectomy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Kazunari Hirota, MD, Kyorin University
Other Study IDs: No.518
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: MicroRNA Expression Profile in Human Vitreous of Various Vitreoretinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3ml of blood serum and 1ml of vitreous
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- human vitreous, human blood serum, PCR: human vitreous and blood serum sampling, PCR
  1ml of human vitreous and 3ml of human blood serum of patients with various vitreoretinal diseases

SUMMARY:
MicroRNAs are important regulators of many cellular functions but their expression profile in human vitreous is still unclear. Aim of this study is to investigate microRNA expression profile by PCR in human vitreous of patients with various vitreoretinal disorders and compare with that of patients with macular holes which are suggested to be similar to that of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* any patients undergoing vitrectomy for various vitreoretinal diseases

Exclusion Criteria:

* previously vitrectomized eyes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pateints undergoing vitrectomy for various vitreoretinal disesases
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MicroRNA expression profile in human vitreous investigated by PCR | 1month

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin University School Of Medicine, Mitakasi Sinkawa6-20-2, Tokyo, Japan